CLINICAL TRIAL: NCT04781322
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Study of Safety, Tolerability, and Bioeffects of Alirocumab in Non-treatment Seeking Heavy Drinkers
Brief Title: Safety, Tolerability, and Bioeffects of Alirocumab in Non-treatment Seeking Heavy Drinkers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10000036; 000036-AA
Record Dates: First submitted 2021-03-03; First posted 2021-03-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-07-25

CONDITIONS: Alcohol Associated Liver Disease; Heavy Drinking Behavior
Keywords: Alcohol; Liver; PCSK9; Fatty Liver; Inflammation
MeSH Terms: conditions — Fatty Liver; Inflammation | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Heavy drinking healthy volunteers
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Heavy drinking healthy volunteers
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alirocumab — Alirocumab is a human monoclonal antibody (IgG1) that binds to and inhibits PCSK9 and was approved by the FDA in July of 2015. PCSK9 binds to and promotes degradation of low-density lipoprotein receptors (LDLR) on hepatocyte membranes.
  Arms: Intervention
Other: Placebo — Heavy drinking healthy volunteers
  Arms: Placebo

SUMMARY:
Background:

Drinking alcohol can lead to swelling and injury in the liver. Long-term heavy drinking may lead to liver disease. Researchers want to study the relationship between a drug called alirocumab, alcohol use, and liver functioning/swelling.

Objective:

To study the effects of alirocumab in people who drink alcohol.

Eligibility:

Healthy adults ages 21 to 65 who regularly consume an average of 20 or more drinks per week.

Design:

Participants will be screened under protocol 14-AA-0181.

Participants will get alirocumab or a placebo as an injection under the skin.

Participants will give blood and urine samples. They will have physical exams.

Participants will have FibroScans . It measures liver and spleen stiffness. Participants will lie on a table. They will expose the lower right and left side of their chest. The machine will send a small vibration to the liver.

Participants may have magnetic resonance imaging (MRI) scans of the liver. The MRI scanner is shaped like a cylinder. Participants will lie on a table that slides in and out of the scanner. A device called a coil will be placed over their liver.

Participants will have a Doppler scan and ultrasound. These tests measure blood flow in the body.

Participants will have an electrocardiogram. It measures heart function.

Participants will fill out surveys about how they are feeling, their alcohol consumption, and other behaviors. They will complete cognitive tasks on a computer.

Participants will meet with a clinician. They will discuss the participant s assessment results, patterns of drinking, and possibly stopping or cutting down on drinking.

Participation will last for 8 weeks. Participants will have 9 study visits.

DETAILED DESCRIPTION:
Study Description:

The PCSK9 inhibitor alirocumab has been recently shown to attenuate alcohol-induced hepatic triglyceride accumulation, hepatocellular injury and hepatic inflammation in a rat model of chronic alcohol exposure. Given the unmet clinical need for novel treatment options for alcohol-associated liver disease (ALD), we are proposing to conduct a safety and tolerability study of alirocumab in this new target population.

We hypothesize that alirocumab will be well tolerated and safe in this new target population and alirocumab will attenuate alcohol-induced liver damage and inflammatory biomarkers.

Objectives:

Primary Objective: The primary objective is to assess the safety and tolerability of alirocumab in subjects who are heavy drinkers.

Secondary/Exploratory Objectives: Secondary/exploratory objectives are to assess various biomarkers related to alcohol-induced liver damage and inflammation.

Endpoints:

Primary Endpoint: The primary endpoint in the study is to assess the incidence and severity of treatment-emergent adverse events in non-treatment seeking heavy drinkers treated with alirocumab or placebo. [Time Frame: baseline to week 8]

Secondary/exploratory Endpoints: The secondary endpoint is to explore effects of alirocumab on various biomarkers using change from baseline.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female between the age of 21 and 65 years.
  2. Ability to provide written informed consent.
  3. Females: Negative urine pregnancy test, not currently breastfeeding, agree to abstain or use accepted form of contraception including use of oral contraceptives; use of barrier method of contraceptive, such as condoms; use of an approved IUD or other long-acting reversible contraceptive (LARC); have a male sexual partner who is surgically sterilized; or have exclusively female sexual partner(s).

     Males: Agree to abstain or use accepted form of contraception, such as condoms.
  4. Current chronic alcohol use, non-treatment seeking heavy drinker (an average of >= 20 standard drinks per week for at least 12 weeks).

EXCLUSION CRITERIA:

1. Treatment seeking for alcohol use disorder.
2. History of a serious hypersensitivity reaction to PCSK9 inhibitors, monoclonal antibodies, or any component of the drug product.
3. Chronic use of statins within eight weeks of the study to treat hypercholesteremia, or fibrates, with the exception of fenofibrates, within six weeks of the study.
4. Current/past use of PCSK9 inhibitors.
5. Clinically significant and/or unstable cardiovascular-disease over the past 12 months.
6. Current or prior history of any clinically significant disease, including, fibromyalgia, severe neuropathic pain, seizure disorder, uncontrolled endocrine disease known to influence serum lipids or lipoproteins, hemorrhagic stroke, cancer within the past 5 years (except for adequately treated basal skin cancer, squamous cell skin cancer, or in situ cervical cancer), uncontrolled (defined as Hgb A1c >8%) or newly diagnosed (within 3 months prior to screening) diabetes, or any other significant abnormality identified at the time of screening that, in the judgment of the investigator or study clinician, would preclude safe completion of the study.
7. Positive HIV test or positive Hepatitis B surface antigen (HBsAg), and/or positive Hepatitis C antibody (HCV) at screening.
8. Alanine aminotransferase or aspartate aminotransferase exceeding 5 times the upper limit of normal levels at screening will be excluded. Bilirubin 2x UNL or Creatinine > 1.5 mg/dl at screening will be excluded.
9. Triglycerides > 400mg/dL (>4.52 mmol/L) at screening.
10. Chronic renal failure as estimated by glomerular filtration rate (GFR) < 60mL/min/1.73 m^2 at screening.
11. Any underlying clinically significant and/or unstable acute or chronic liver disease unrelated to alcohol use at screening.
12. Patients with coagulopathy defined as INR >1.5, prothrombin time prolonged by > 3s, and/or platelets <75,000 / mm^3 at screening.
13. Use of any medications that interfere with blood clotting.
14. Patients with significant hematologic abnormalities.
15. Significant obesity (Obesity Class III) defined as BMI greater than or equal to 40 at screening.
16. History of previous bariatric surgery or transplant surgery.
17. History of plasmapheresis treatment within 2 months prior to screening or plans to undergo plasmapheresis during the study.
18. Use of the following medications: Any medication that requires intramuscular administration injections. Systemic corticosteroids, unless used as replacement therapy for pituitary/adrenal disease with a stable regimen for at least 6 weeks prior to screening. Estrogen or testosterone therapy, unless regimen stable for 6 weeks prior to screening visit.
19. Use of any investigational drugs within 1 month, or five half-lives, whichever is longer, of the study procedures.
20. Plan to use red yeast rice during the study.
21. Presence of any current suicidality.
22. History of epilepsy or alcohol-related seizures in the last 12 months.
23. Any other severe condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study, such as psychosis, delirium or acute change of mental status.

For optional MRI: a) Presence of ferromagnetic objects in the body that may be adversely affected by or contraindicated for MRI, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report b) Use of MRI-incompatible intrauterine device (IUD).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the safety and tolerability of alirocumab in subjects who are heavy drinkers. | 8 weeks
  The primary endpoint in the study is to assess the incidence and severity of treatment-emergent adverse events in non-treatment seeking heavy drinkers treated with alirocumab or placebo.

SECONDARY OUTCOMES:
Secondary/exploratory objectives are to assess various biomarkers related to alcohol-induced liver damage and inflammation. | ongoing
  These biomarkers will assess various biological processed in AUD, such as inflammation, liver biology and clinical alcohol-related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Falk W Lohoff, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000036-AA.html